CLINICAL TRIAL: NCT05109403
Title: Comparison of Ovarian Response in Oocyte Donors Triggered With GnRH Agonists Depending on the LH Level the Day After the Triggering
Brief Title: Ovarian Response in Oocyte Donors Triggered With GnRH Agonists
Status: Completed | Type: Observational
Sponsor: Clínica EUGIN (Other)
Responsible Party: Sponsor
Other Study IDs: AGOTRIG
Record Dates: First submitted 2021-10-27; First posted 2021-11-05 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-03

CONDITIONS: Poor Response to Ovulation Induction
Keywords: oocyte donation; agonist ovulation trigger

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- LH post-trigger < 15 UI/l: Oocyte donors that present with LH levels < 15UI/I, post trigger by agonists of GnRH
- LH post-trigger > 15 UI/l: Oocyte donors that present with LH levels > 15UI/I, post trigger by agonists of GnRH

SUMMARY:
The use of agonist of GnRH (aGnRH) trigger to avoid ovarian hyperstimulation syndrome is nowadays widely used. The action of the aGnRH in the hypophysis triggers an LH and FSH surge, which mimicks the natural surge that occurs in the middle of a natural cycle, and thus being able to elicit the ovulation. However, in some patients the aGnRH trigger ends in a poor oocyte recuperation, and that has led some physicians to measure the LH surge after the aGnRH trigger to check its effectiveness.

Even though there is still some discrepancy about the exact cut-off value for a proper LH surge 12h after the aGnRH trigger, most of the published papers report the value of 15UI/L as an adequate threshold under which the results of the pick-up are suboptimal. Other authors even report a value of 52UI/L to predict a decrease in oocyte retrieval and maturity rate and a value of 15UI/L to predict a dramatic decrease in the results.

Some of the abovementioned studies report that the basal LH value or the LH value on the day of the trigger could also be predictive of suboptimal responses. Additionally, some authors have tried to "rescue" the suboptimal patients with a retrigger of hCG, or they have compared those suboptimal responders with patients triggered with both aGnRH and low doses of hCG. In both cases the addition of hCG seems to improve the results.

Most of the scientific bibliography available so far is based on infertile patients undergoing IVF treatments, while in some papers both IVF patients and egg donors have been analyzed. The current study involves exclusively oocyte donation cycles, where the final aim is to identify donors at a high risk of a suboptimal response, and to potentially improve results by potentially adding low doses of hCG (1000 UI).

ELIGIBILITY:
Inclusion Criteria:

* Oocyte donors included in the oocyte donation program of Clinica EUGIN that have been triggered with GnRH agonists.
* Any cycle of oocyte donation from the program of Clinica EUGIN, regardless of the type and dose of gonadotropin used for stimulation.

Exclusion Criteria:

- None.

Ages: 18 Years to 34 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: Oocyte donors included in the oocyte donation program of Clinica EUGIN
Sampling Method: Non-Probability Sample
Enrollment: 224 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-01-26 (Actual); Study Completion 2022-02-10 (Actual)

PRIMARY OUTCOMES:
Oocyte retrieval rate | 30 days
  Number of cumulus oocyte complexes (COCs) retrieved divided by the number of follicles > 14mm the day of the last follicular control

SECONDARY OUTCOMES:
Oocyte maturity rate | 30 days
  Number of metaphase-II mature oocytes retrieved divided by the number of COCs retrieved

CONTACTS AND LOCATIONS:
Overall Officials: Anna Blázquez Ventura, MD, PhD, Principal Investigator — Clinica EUGIN
Locations (1):
- Clinica EUGIN, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Blazquez A, Falco N, Cano E, Rodriguez F, Vassena R, Miguel-Escalada I, Popovic M, Rodriguez A. No association between LH levels and ovarian response in oocyte donors triggered with gonadotropin-releasing hormone agonist: A prospective study. Eur J Obstet Gynecol Reprod Biol. 2024 Mar;294:163-169. doi: 10.1016/j.ejogrb.2024.01.022. Epub 2024 Jan 18. PMID 38266482